CLINICAL TRIAL: NCT02316847
Title: Multi-center, Open-label, Study of Safety and Tolerability of Chronic Intermittent Usage of Diazepam Nasal Spray in Adolescents and Adult Patients With Cluster Seizures, Including Assessment of Olfaction and Reported Changes in Taste.
Brief Title: An Open-Label, Safety and Tolerability Study of Chronic Intermittent Use of Diazepam Nasal Spray.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZNS-EP-1025
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy
Keywords: Cluster Seizures; Seizures; Clusters; Acute repetitive seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diazepam nasal spray (Adults) (Experimental): One dose of diazepam nasal spray is two intranasal sprays; one in each nostril using a nasal spray device. The dose is administered while the subject is sitting up or lying down.
  Interventions: Drug: diazepam nasal spray
- Diazepam Nasal Spray (Adolescents) (Experimental): One dose of diazepam nasal spray is two intranasal sprays; one in each nostril using a nasal spray device. The dose is administered while the subject is sitting up or lying down.
  Interventions: Drug: diazepam nasal spray

INTERVENTIONS:
Drug: diazepam nasal spray

SUMMARY:
This study will assess long-term safety and tolerability of repeat dose diazepam nasal spray in adolescents and adults with cluster seizures, with a focus on potential local effects (changes in nasal mucosa, olfaction, and taste).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of drug-resistant epilepsy
* Patients who experience multiple episodes of acute repetitive seizures requiring at least one concomitant antiepileptic drug (AED)
* Occurrence of at least 3 seizure clusters within the past 12 months, including at least one cluster in the 4 months prior to the Screening Visit
* A caregiver must consent to participate together with the subject for purposes of observation and data collection
* The caregiver must be present when the investigational product is administered
* Screening body weight between 26 to 111 kg, inclusive

Exclusion Criteria:

* Female subject who is pregnant, breastfeeding, or planning to become pregnant
* Presence or history of any abnormality or illness that may affect the absorption, distribution, metabolism or elimination of diazepam
* Known allergy or hypersensitivity to diazepam, related drugs, or any of the formulation components
* Positive screening test for ethanol or other drugs of abuse
* Unable to receive medications intranasally

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MinJae Lee, Study Director — SK Biopharmaceuticals Co, Ltd
Locations (33):
- United States (33):
  - Acorda Site #227, Phoenix, Arizona
  - Acorda Site #204, Little Rock, Arkansas
  - Acorda Site #213, Los Angeles, California
  - Acorda Site #220, Orange, California
  - Acorda Site #206, Orlando, Florida
  - Acorda Site #241, Port Charlotte, Florida
  - Acorda Site #231, Tallahassee, Florida
  - Acorda Site #201, Tampa, Florida
  - Acorda Site #234, Tampa, Florida
  - Acorda Site #217, Augusta, Georgia
  - Acorda Site #232, Honolulu, Hawaii
  - Acorda Site #225, Fort Wayne, Indiana
  - Acorda Site #226, Ames, Iowa
  - Acorda Site #202, Bethesda, Maryland
  - Acorda Site #212, Boston, Massachusetts
  - Acorda Site #214, Boston, Massachusetts
  - Acorda Site #208, Boston, Massachusetts
  - Acorda Site #216, Kansas City, Missouri
  - Acorda Site #205, St Louis, Missouri
  - Acorda Site #222, Hackensack, New Jersey
  - Acorda Site #223, New York, New York
  - Acorda Site #233, Rochester, New York
  - Acorda Site #230, Portland, Oregon
  - Acorda Site #219, Philadelphia, Pennsylvania
  - Acorda Site #237, Philadelphia, Pennsylvania
  - Acorda Site #203, Charleston, South Carolina
  - Acorda Site #235, Memphis, Tennessee
  - Acorda Site #218, Nashville, Tennessee
  - Acorda Site #221, Dallas, Texas
  - Acorda Site #229, Houston, Texas
  - Acorda Site #215, Richmond, Virginia
  - Acorda Site #224, Renton, Washington
  - Acorda Site #210, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents or adults who have refractory epilepsy (drug resistant epilepsy per Kwan 2010) with a history of cluster seizures, also known as multiple episodes of acute repetitive seizures, for which acute treatment with a benzodiazepine was indicated as part of the standard of care or an individualized rescue treatment plan.
Groups:
- DZNS - Adolescents (Ages 12 - 15); DZNS - Adults (Ages 16 - 65): One dose of diazepam nasal spray is two intranasal sprays; one in each nostril using a nasal spray device. The dose is administered while the subject is sitting up or lying down.
Period: Overall Study
Arm/Group | DZNS - Adolescents (Ages 12 - 15) | DZNS - Adults (Ages 16 - 65)
Started | 9 | 99
Completed | 0 | 13
Not Completed | 9 | 86
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 9
Not completed — Noncompliance with study drug | 0 | 3
Not completed — Withdrawn due to termination by Sponsor | 7 | 67

BASELINE CHARACTERISTICS:
Groups:
- Diazapam Nasal Spray (DZNS) Adults; Diazapam Nasal Spray (DZNS) Adolescents: One dose of diazepam nasal spray is two intranasal sprays; one in each nostril using a nasal spray device. The dose is administered while the subject is sitting up or lying down.
- Total: Total of all reporting groups
Arm/Group | Diazapam Nasal Spray (DZNS) Adults | Diazapam Nasal Spray (DZNS) Adolescents | Total
Number analyzed (Participants) | 99 | 9 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 9 | 16
  Between 18 and 65 years | 91 | 0 | 91
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (12.58) | 13.4 (1.13) | 32.9 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 3 | 51
  Male | 51 | 6 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 93 | 7 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 5 | 0 | 5
  Black or African American | 9 | 1 | 10
  White | 75 | 8 | 83
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 7 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 9 | 108

OUTCOME MEASURES:

1. Primary Outcome: Olfactory Changes as Measured by the Smell Identification Test (SIT)
Description: The SIT is a 50-item multiple-choice standardized test of olfactory function. Scoring of the test in the ability to smell ranges from normal (Normosmia: score 35 - 40 Women; 34 - 40 Men); to inability to smell (Anosmia score 6 - 18); or Malingering (not engaged in the test) ranges 0 - 5.
Time Frame: Screening, weeks 12, 24, 36, 48 and 51
Population: Of 91 subjects in the Safety Population, data was available for 62 subjects at screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Diazepam Nasal Spray (Adults) | Diazepam Nasal Spray (Adolescents)
Number analyzed (Participants) | 57 | 5
Participants
  Screening: Normosmia | 18 | 0
  Screening: Mild Microsmia | 15 | 1
  Screening: Moderate Microsmia | 8 | 3
  Screening: Severe Micromisia | 7 | 1
  Screening: Anosmia | 9 | 0
  Screening: Probable Malingering | 0 | 0
  Week 12: number analyzed (Participants) | 34 | 3
  Week 12: Normosmia | 6 | 0
  Week 12: Mild Microsmia | 16 | 0
  Week 12: Moderate Microsmia | 9 | 1
  Week 12: Severe Micromisia | 1 | 2
  Week 12: Anosmia | 2 | 0
  Week 12: Probable Malingering | 0 | 0
  Week 24: number analyzed (Participants) | 21 | 0
  Week 24: Normosmia | 5 | 0
  Week 24: Mild Microsmia | 9 | 0
  Week 24: Moderate Microsmia | 2 | 0
  Week 24: Severe Micromisia | 5 | 0
  Week 24: Anosmia | 0 | 0
  Week 24: Probable Malingering | 0 | 0
  Week 36: number analyzed (Participants) | 14 | 0
  Week 36: Normosmia | 2 | 0
  Week 36: Mild Microsmia | 6 | 0
  Week 36: Moderate Microsmia | 4 | 0
  Week 36: Severe Micromisia | 1 | 0
  Week 36: Anosmia | 1 | 0
  Week 36: Probable Malingering | 0 | 0
  Week 48: number analyzed (Participants) | 10 | 0
  Week 48: Normosmia | 0 | 0
  Week 48: Mild Microsmia | 5 | 0
  Week 48: Moderate Microsmia | 1 | 0
  Week 48: Severe Micromisia | 3 | 0
  Week 48: Anosmia | 1 | 0
  Week 48: Probable Malingering | 0 | 0
  Week 51: number analyzed (Participants) | 10 | 0
  Week 51: Normosmia | 1 | 0
  Week 51: Mild Microsmia | 3 | 0
  Week 51: Moderate Microsmia | 1 | 0
  Week 51: Severe Micromisia | 4 | 0
  Week 51: Anosmia | 1 | 0
  Week 51: Probable Malingering | 0 | 0

2. Primary Outcome: Change From Baseline (Screening) in Nasal Mucosa.
Description: Change from baseline treatment visits using a focused nasal exam was based on a scale of nasal irritation "none" to Grade 4 "septal perforation."
Time Frame: Screening, Weeks 12, 24, 36, 48 and 51
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Adults; Adolescents: One dose of diazepam nasal spray is two intranasal sprays; one in each nostril using a nasal spray device. The dose is administered while the subject is sitting up or lying down.
Arm/Group | Adults | Adolescents
Number analyzed (Participants) | 84 | 7
Participants
  Screening : Nasal Irritation None | 67 | 6
  Screening : Nasal Irritation Grade 1a | 10 | 1
  Screening : Nasal Irritation Grade 1b | 3 | 0
  Screening : Nasal Irritation Grade 2 | 0 | 0
  Screening : Mucosal Edema None | 71 | 6
  Screening : Mucosal Edema Mild | 9 | 1
  Screening : Nasal Discharge None | 66 | 6
  Screening : Nasal Discharge Mild | 14 | 1
  Screening : Mucosal Erythema None | 65 | 5
  Screening : Mucosal Erythema Mild | 13 | 2
  Screening : Mucosal Erythema Moderate | 2 | 0
  Screening : Mucosal Bleeding/Epistaxis None | 79 | 6
  Screening : Mucosal Bleeding/Epistaxis Mild | 1 | 1
  Screening : Crusting of Mucosa None | 77 | 7
  Screening : Crusting of Mucosa Mild | 3 | 0
  Week 12 : Nasal Irritation None | 50 | 4
  Week 12 : Nasal Irritation Grade 1a | 5 | 0
  Week 12 : Nasal Irritation Grade 1b | 3 | 0
  Week 12 : Nasal Irritation Grade 2 | 1 | 0
  Week 12 : Mucosal Edema None | 55 | 3
  Week 12 : Mucosal Edema Mild | 4 | 1
  Week 12 : Nasal Discharge None | 49 | 4
  Week 12 : Nasal Discharge Mild | 10 | 0
  Week 12 : Mucosal Erythema None | 39 | 4
  Week 12 : Mucosal Erythema Mild | 20 | 0
  Week 12 : Mucosal Erythema Moderate | 0 | 0
  Week 12 : Mucosal Bleeding/Epistaxis None | 58 | 4
  Week 12 : Mucosal Bleeding/Epistaxis Mild | 1 | 0
  Week 12 : Crusting of Mucosa None | 58 | 4
  Week 12 : Crusting of Mucosa Mild | 1 | 0
  Week 24: Nasal Irritation None | 37 | 1
  Week 24: Nasal Irritation Grade 1a | 1 | 0
  Week 24: Nasal Irritation Grade 1b | 1 | 0
  Week 24: Mucosal Edema None | 35 | 0
  Week 24: Mucosal Edema Mild | 4 | 1
  Week 24: Nasal Discharge None | 31 | 1
  Week 24: Nasal Discharge Mild | 8 | 0
  Week 24: Mucosal Erythema None | 33 | 1
  Week 24: Mucosal Erythema Mild | 6 | 0
  Week 24: Mucosal Bleeding/Epistaxis None | 39 | 1
  Week 24: Crusting of Mucosa None | 37 | 1
  Week 24: Crusting of Mucosa Mild | 2 | 0
  Week 36: Nasal Irritation None | 21 | 1
  Week 36: Nasal Irritation Grade 1a | 1 | 0
  Week 36: Mucosal Edema None | 21 | 0
  Week 36: Mucosal Edema Mild | 1 | 1
  Week 36: Nasal Discharge None | 20 | 1
  Week 36: Nasal Discharge Mild | 1 | 0
  Week 36: Mucosal Erythema None | 20 | 1
  Week 36: Mucosal Erythema Mild | 2 | 0
  Week 36: Mucosal Bleeding/Epistaxis None | 22 | 1
  Week 36: Crusting of Mucosa None | 21 | 1
  Week 36: Crusting of Mucosa Mild | 1 | 0
  Week 48: Nasal Irritation None | 12 | 0
  Week 48: Nasal Irritation Grade 1a | 1 | 0
  Week 48: Mucosal Edema None | 13 | 0
  Week 48: Nasal Discharge None | 13 | 0
  Week 48: Mucosal Erythema None | 13 | 0
  Week 48: Mucosal Bleeding/Epistaxis None | 13 | 0
  Week 48: Crusting of Mucosa None | 13 | 0
  Week 51: Nasal Irritation None | 13 | 0
  Week 51: Mucosal Edema None | 13 | 0
  Week 51: Nasal Discharge None | 12 | 0
  Week 51: Nasal Discharge Mild | 1 | 0
  Week 51: Mucosal Erythema None | 13 | 0
  Week 51: Mucosal Bleeding/Epistaxis None | 13 | 0
  Week 51: Crusting of Mucosa None | 13 | 0

3. Primary Outcome: Change in Taste as Measured by a Taste Change Questionnaire
Description: Change in taste questionnaire was administered to subjects at every study visit only if the subject complained of a change in taste or as needed to report a related AE. The taste change profile included sweet, salty, sour, bitter, oily, sharp, chalky, metallic. The subject rated the change on a 10-point scale ranging from a weak change (1) to very strong (10).
Time Frame: Weeks 12, 24
Population: Safety Population - Number of subjects with at least one change in taste after dose administration. 6 Adults at 12 Weeks and 4 Adults at 24 weeks. No Adolescents participated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diazepam Nasal Spray (Adults)
Number analyzed (Participants) | 84
units on a scale
  Week 12: number analyzed (Participants) | 6
  Week 12 | 7.7 (2.73)
  Week 24: number analyzed (Participants) | 4
  Week 24 | 8.3 (0.50)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reported on the safety population which included only those who received at least one dose of DZNS. Adults = 84 Adolescents = 7
Arm/Group | Adults | Adolescents
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/7
Serious Adverse Events (participants affected / at risk) | 11/84 | 1/7
Other Adverse Events (participants affected / at risk) | 64/84 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (N=84) | Adolescents (N=7)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Oesophagitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diebetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 2 | 0
Status Epilepticus (Nervous system disorders) | 3 | 1
Status Migrainosus (Nervous system disorders) | 1 | 0
Psychogenic Seizure (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (N=84) | Adolescents (N=7)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 25 | 2
Dysgeusia (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Overdose (Injury, poisoning and procedural complications) | 6 | 0
Lacrimation increased (Eye disorders) | 7 | 1
Somnolence (Nervous system disorders) | 6 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.